CLINICAL TRIAL: NCT02537509
Title: Multicentre, Cross-over, PRAgmatic Trial in Atopic Dermatitis Testing Long-term Control Effectiveness of New Phototherapy Regimen During Winter as an add-on Therapy, Coupled With Oral Vitamin D Supplementation vs. Placebo in a Randomised, Parallel-group Trial
Brief Title: PRAgmatic Trial in Atopic Dermatitis Testing Long-term Control Effectiveness of New Phototherapy Regimen During Winter Coupled With Oral Vitamin D Supplementation vs. Placebo
Acronym: PRADA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-000881-73; 35RC14_9754_PRADA (Other: CHU de Rennes)
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecalciferol (Active Comparator): Administration of cholecalciferol every 3 months during 2 years combined with new phototherapy regimen during winter (phototherapy winter 1, observation winter 2 or the opposite)
  Interventions: Drug: Cholecalciferol
- Placebo of cholecalciferol (Placebo Comparator): Administration of placebo of cholecalciferol every 3 months during 2 years combined with new phototherapy regimen during winter (phototherapy winter 1, observation winter 2 or the opposite)
  Interventions: Drug: Placebo of cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol
  Other Names: Uvedose
  Arms: Cholecalciferol
Drug: Placebo of cholecalciferol
  Other Names: Placebo of Uvedose
  Arms: Placebo of cholecalciferol

SUMMARY:
Spaced phototherapy sessions during winter as add-on therapy in combination with vitamin D supplementation or not, could be beneficial to improve disease LTC in AD patients

DETAILED DESCRIPTION:
The major therapeutic challenge in patient with Atopic Dermatitis is long-term control of disease activity (LTC), for which the current TAT-based pro-active strategy does not meet all the needs.

Phototherapy is a good candidate: it is widely used as a second-line treatment in AD with demonstrated efficacy. However, only short-term control has been evaluated; and only 2-3 times a week intensive schedules have been tested and are used in current practice. A novel phototherapy regimen would be required for disease LTC, allowing a trade-off between disease control, UV-induced risks, and patient adherence.

Vitamin D supplementation is another good candidate: several studies have shown lower serum levels of vitamin D to be correlated with more severe AD; and three short-term, low-power low-quality, placebo-controlled randomised trials testing vitamin D supplementation yielded conflicting results, leaving its therapeutic efficacy undecided for short-term control, and unknown for LTC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atopic dermatitis (Hanifin and Rajka criteria),
* Aged 15 years or more,
* With > 2 years of disease evolution,
* With moderate-to-severe disease (IGA > 2),
* Patients that have received TAT for at least 12 weeks and have symptoms requiring an increase in therapy,
* Seasonality in disease severity (based on a questionnaire assessing disease improvement during summer),
* Easy access to a phototherapy cabin (widely implanted in primary care dermatology private practice in France),
* Effective contraception to be used at least 30 days before initiation of treatment, during treatment and 29 weeks after last administration for women of reproductive age,
* Written informed consent of the patient
* For patients aged between 15 and 18, written informed consent of the parents and of the teenager.

Exclusion Criteria:

* Any cause of contra-indication for vitamin D supplementation: flare of granulomatosis, primary hyperparathyroidism,
* Clinical suspicion of hypercalciuria,
* Indication to a systemic immunosuppressant in the next 2 years,
* Atopic dermatitis known to be aggravated by UV exposure,
* Any contra-indication for artificial or solar exposure including: genetic diseases with a predisposition to skin cancer, any history of personal skin cancer (melanoma, squamous cell skin cancer, basal cell skin cancer), lupus, dermatomyositis, any other photosensitizing skin disease, photosensitizing medication (see appendix 2),
* More than 100 previous phototherapy sessions in lifetime,
* Pregnancy or breastfeeding,
* Persons subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Hierarchical criterion based on repeated measures of PO-SCORAD severity score | 2 years
  Measurement of PO-SCORAD score
Hierarchical criterion based on cumulative consumption of topical anti-inflammatory treatments (collected tubes) during winter | 2 years
  Measurement of cumulative consumption of topical anti-inflammatory treatments

SECONDARY OUTCOMES:
Assessment of desease severity | 2 years
  Assessment of desease severity by EASI score
Assessment of desease severity | 2 years
  Assessment of desease severity by IGA score
Assessment of desease severity | 2 years
  Assessment of desease severity by SCORAD score
Assessment of desease severity | 2 years
  Assessment of desease severity by POEM score
Assessment of the quality of life | 2 years
  Assessment of the quality of life by DLQI score
Measurement of serum Vitamin D (25-(OH)-vitamin D) | 2 years
Measurement of total IgE serum | 2 years
Assessement of number of weeks of well-controlled atopic dermatitis | 2 years
Assessment of inter-visit cumulative consumption of topical anti-inflammatory treatments | 2 years
Assessment of patient satisfaction | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Droitcourt, Principal Investigator — Rennes University Hospital
Locations (11):
- France (11):
  - Hôpital Saint André, Bordeaux
  - Hôpital Morvan, Brest
  - Hôpital Trousseau, Chambray-lès-Tours
  - Centre Hospitalier, Le Mans
  - CHU de Nantes - Hôtel Dieu, Nantes
  - APHP - Hôpital Tenon, Paris
  - Centre Hospitalier, Périgueux
  - Hôpital Laënnec, Quimper
  - Hôpital Pontchaillou, Rennes
  - CHR St Brieuc, Saint-Brieuc
  - Centre Hospitalier, Valenciennes

REFERENCES:
- [Derived] Droitcourt C, Barbarot S, Maruani A, Darrieux L, Misery L, Brenaut E, Adamski H, Chabbert C, Vermersch A, Weiborn M, Seneschal J, Taieb A, Plantin P, Maillard H, Phan A, Skowron F, Viguier M, Staumont-Salle D, Nosbaum A, Soria A, Barbaud A, Oger E, Dupuy A; Groupe de Recherche sur l'Eczema Atopique de la Societe Francaise de Dermatologie (GREAT). A new phototherapy regimen during winter as an add-on therapy, coupled with oral vitamin D supplementation, for the long-term control of atopic dermatitis: study protocol for a multicentre, randomized, crossover, pragmatic trial - the PRADA trial. Trials. 2019 Mar 25;20(1):184. doi: 10.1186/s13063-019-3276-9. PMID 30909923